CLINICAL TRIAL: NCT00041808
Title: A Phase I/II Single Dose Trial to Determine The Safety, Tolerance, Pharmacokinetic Profile, and Preliminary Activity of Intrahepatic Delivery (Via Hepatic Artery Catheterization) of Doxorubicin Hydrochloride Adsorbed to Magnetic Targeted Carriers ( MTC-DOX) in Patients With Metastatic Cancer to the Liver .
Brief Title: Magnetic-Targeted Doxorubicin in Treating Patients With Cancer Metastatic to the Liver
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: FeRx (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTC-DOX-003; NCT00023803 (obsolete NCT alias)
Record Dates: First submitted 2002-07-17; First posted 2002-07-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-02

CONDITIONS: Metastases, Neoplasm; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Breast Neoplasms; Melanoma; Sarcoma; Gastrointestinal Neoplasms; Lung Neoplasms; Liver Neoplasms; Cholangiocarcinoma
Keywords: Metastatic liver cancer; Cholangiocarcinoma; colorectal cancer; esophageal cancer; gastric cancer; pancreatic cancer; breast cancer; malignant melanoma; sarcoma; GIST; gastrointestinal stromal tumor; lung cancer; liver cancer
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Breast Neoplasms; Melanoma; Sarcoma; Gastrointestinal Neoplasms; Lung Neoplasms; Liver Neoplasms; Cholangiocarcinoma; Gastrointestinal Stromal Tumors | interventions — Injections; Drug Therapy

INTERVENTIONS:
Drug: MTC-DOX for Injection
Procedure: Chemotherapy

SUMMARY:
MTC-DOX is Doxorubicin or DOX, a chemotherapy drug, that is adsorbed, or made to "stick", to magnetic beads (MTCs). MTCs are tiny, microscopic particles of iron and carbon. When DOX is added to MTCs, DOX attaches to the carbon part of the MTCs. MTC-DOX is directed to and deposited in the area of a tumor, where it is thought that it then "leaks" through the blood vessel walls. Once in the surrounding tissues, it is thought that Doxorubicin becomes "free from" the magnetic beads and will then be able to act against the tumor cells. The iron component of the particle has magnetic properties, making it possible to direct MTC-DOX to specific tumor sites in the liver by placing a magnet on the body surface. It is hoped that MTC-DOX used with the magnet may target the chemotherapy drug directly to liver tumors and provide a treatment to patients with cancers that have spread to the liver.

ELIGIBILITY:
Inclusion Criteria

* Patients with a Karnofsky (or equivalent) performance status > 60 and an expected survival of > 2 months
* Patients agreeing to use a medically effective method of contraception
* Patients able to understand and give written informed consent
* The center of the tumor mass must be < or = 14 cm from the anterior or lateral abdominal wall as determined by cross sectional imaging measured at baseline. This is required for optimal retention of MTC-DOX by the magnetic field. If more than one tumor mass is present, all of the treated tumor masses must meet this criterion

Exclusion Criteria

* Women who are pregnant or lactating
* Patient's with metastatic liver cancer, or other primary liver cancer excluding HCC, with diffuse disease that does not have focal area(s) conducive to local regional therapy
* Patients with the following laboratory abnormalities:Hemoglobin < 10.0 g/dL;Granulocyte count < 1,500 per mm3;Platelet count < 50,000 per mm3; Lymphocyte count < 0.5 x 10 to the 9th per L; Total bilirubin >/= 3.0 mg/dL;AST or ALT >/= 5x the upper limit of normal;INR >/= 1.3; Creatinine >/= 2.0 mg/dL
* Patients with either significant cardiovascular disease or any other organ system dysfunction which, in the opinion of the investigator, would either compromise the patient's safety or interfere with the evaluation of the test material. Patients with evidence of a myocardial infarction within six (6) months prior to this trial will be excluded.
* Patients with an indwelling cardiac pacemaker, cerebral aneurysm clips, or any other indwelling device or appliance that could be adversely affected by the use of the external magnet
* Patients at the time of study entry with a second invasive cancer other than basal cell and squamous cell carcinoma of the skin, or carcinoma in situ of the cervix
* Patients with documented evidence of hemachromatosis or hemosiderosis
* Patients with CT or ultrasound evidence of portal vein invasion or thrombosis
* Patients who have had prior anthracycline therapy with a left ventricular ejection fraction (LVEF) <50%, as measured by either multigated radionuclide angiography (MUGA) scan or echocardiogram.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-07; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Joy Koda, PhD, Study Chair
Locations (4):
- United States (3):
  - Scripps Stevens Cancer Division, San Diego, California
  - UCSF Cancer Center, San Francisco, California
  - Scott and White Clinic, Temple, Texas
- Frankfurt Universtiy, Frankfurt, Germany